CLINICAL TRIAL: NCT05227690
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Efficacy, Safety, and Tolerability of Two Fixed Doses (10 mg and 30 mg QD) of CVL-231 (Emraclidine) in Participants With Schizophrenia Experiencing an Acute Exacerbation of Psychosis
Brief Title: A Trial of 10 and 30 mg Doses of CVL-231 (Emraclidine) in Participants With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVL-231-2001; 2022-000580-52 (EudraCT Number)
Record Dates: First submitted 2022-01-27; First posted 2022-02-07 (Actual); Results first posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Schizophrenia Spectrum and Other Psychotic Disorders; Mental Disorders
MeSH Terms: conditions — Schizophrenia; Schizophrenia Spectrum and Other Psychotic Disorders; Mental Disorders

STUDY DESIGN:
Intervention Model Description: Placebo-controlled
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants received placebo tablets orally once daily (QD) through Day 45 of Week 6.
  Interventions: Drug: Placebo
- Emraclidine 10 mg, once daily (QD) (Experimental): Participants received emraclidine 10 mg tablets orally once daily (QD) through Day 45 of Week 6.
  Interventions: Drug: Emraclidine 10 mg
- Emraclidine 30 mg, once daily (QD) (Experimental): Participants received emraclidine 30 mg tablets orally once daily (QD) through Day 45 of Week 6.
  Interventions: Drug: Emraclidine 30 mg

INTERVENTIONS:
Drug: Placebo — Matching placebo, oral (tablet), once per day for 6 weeks
  Arms: Placebo
Drug: Emraclidine 10 mg — Emraclidine 10 mg, oral (tablet), once per day for 6 weeks
  Other Names: CVL-231; ABBV-1231
  Arms: Emraclidine 10 mg, once daily (QD)
Drug: Emraclidine 30 mg — Emraclidine 30 mg, oral (tablet), once per day for 6 weeks
  Other Names: CVL-231; ABBV-1231
  Arms: Emraclidine 30 mg, once daily (QD)

SUMMARY:
This is a Phase 2, multicenter, randomized, double-blind, placebo-controlled, parallel-group, 6-week trial to evaluate the efficacy, safety, and tolerability of 2 fixed doses of CVL-231 (Emraclidine) (10 mg QD and 30 mg QD) in male and female participants who have schizophrenia and are experiencing an acute exacerbation of psychosis.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of schizophrenia per DSM-5, as confirmed by the MINI for Psychotic Disorders.
* CGI-S ≥4 (moderately to severely ill) at the time of signing the ICF and Baseline.
* PANSS Total Score between 85 and 120, inclusive, at the time of signing the ICF and at Baseline.
* Experiencing an acute exacerbation or relapse of psychotic symptoms, with onset less than 60 days prior to signing the ICF.
* Willing to discontinue all prohibited medications to meet protocol-required washouts prior to and during the trial period.
* Body mass index of 18.0 to 40.0 kg/m2 and a total body weight ≥50 kg (110 lbs).
* Ability, in the opinion of the investigator, to understand the nature of the trial, participate in trial visits, and comply with protocol requirements.

Exclusion Criteria:

* Current DSM-5 diagnosis other than schizophrenia (note: anxiety symptoms secondary to schizophrenia are allowed); Acute depressive symptoms within 30 days prior to signing the ICF that require treatment with an antidepressant are exclusory. Acute manic symptoms within 30 days prior to signing the ICF that require treatment with a mood stabilizer are exclusory.
* Any of the following:

  * Schizophrenia considered resistant/refractory to antipsychotic treatment by history (failure to respond to 2 or more courses of adequate pharmacological treatment defined as an adequate dose per label and a treatment duration of at least 4 weeks)
  * History of response to clozapine treatment only or failure to respond to clozapine treatment
* Any of the following regarding history of schizophrenia:

  * Time from initial onset of schizophrenia <2 years based on prior records or participant self-report
  * Presenting with an initial diagnosis of schizophrenia
  * Presenting for the first time with an acute psychotic episode requiring treatment
* Reduction (improvement) in PANSS total score of ≥20% between Screening and Baseline.
* Current or past history of significant cardiovascular, pulmonary, gastrointestinal, renal, hepatic, metabolic, genitourinary, endocrine (including diabetes mellitus), malignancy (except for basal cell carcinoma of the skin and cervical carcinoma in situ, at the discretion of the investigator), hematological, immunological, neurological, or psychiatric disease that, in the opinion of the investigator or medical monitor, could compromise either participant safety or the results of the trial.
* Active central nervous system infection, demyelinating disease, degenerative neurological disease, brain tumor, prior hospitalization for severe head trauma, seizures (excluding febrile seizures in childhood), or any central nervous system disease deemed to be progressive during the course of the trial that may confound the interpretation of the trial results
* Diagnosis of moderate to severe substance or alcohol-use disorder (excluding nicotine or caffeine) as per DSM-5 criteria within 12 months prior to signing the ICF.
* Risk for suicidal behavior as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS) and investigator's clinical assessment.
* Any condition that could possibly affect drug absorption.
* Use of prohibited medications prior to randomization within the required wash-out period or likely to require prohibited concomitant therapy during the trial.
* Clinically significant abnormal findings on the physical examination, medical history review, ECG, or clinical laboratory results at screening.
* Positive pregnancy test result prior to receiving IMP. Note: female participants who are pregnant, breastfeeding, or planning to become pregnant during IMP treatment or within 7 days after the last dose of IMP are also excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2024-08-23 (Actual); Study Completion 2024-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (25):
- United States (21):
  - Little Rock, Arkansas, Little Rock, Arkansas
  - Anaheim, California, Anaheim, California
  - Garden Grove, California, Garden Grove, California
  - Lemon Grove, California, Lemon Grove, California
  - Montclair, California, Montclair, California
  - Riverside, California, Riverside, California
  - San Diego, California, San Diego, California
  - Hialeah, Florida, Hialeah, Florida
  - Hollywood, Florida, Hollywood, Florida
  - Mangonia Park, Florida, Mangonia Park, Florida
  - Oakland Park, Florida, Oakland Park, Florida
  - Atlanta, Georgia, Atlanta, Georgia
  - Decatur, Georgia, Decatur, Georgia
  - Shreveport, Louisiana, Shreveport, Louisiana
  - Gaithersburg, Maryland, Gaithersburg, Maryland
  - Flowood, Mississippi, Flowood, Mississippi
  - North Canton, Ohio, North Canton, Ohio
  - DeSoto, Texas, DeSoto, Texas
  - Houston, Texas, Houston, Texas
  - Irving, Texas, Irving, Texas
  - Richardson, Texas, Richardson, Texas
- Bulgaria (4):
  - Stara Zagora, Stara Zagora
  - Veliko Tarnovo, Veliko Tarnovo
  - Veliko Tarnovo, Veliko Tarnovo, Veliko Tarnovo
  - Vratsa, Vratsa, Vratsa

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted at 23 sites in the United States and Bulgaria.
Pre-assignment Details: The study included an up to 15-day Screening Period, 45-day Inpatient Treatment Period, and 28-day Follow-up Period. Participants were randomized in a 1:1:1 ratio to 1 of 3 treatment groups (emraclidine 10 mg QD, emraclidine 30 mg QD, or placebo QD), with randomization stratified by geographic region (United States or all other countries).
Period: Overall Study
Arm/Group | Placebo | Emraclidine 10 mg, Once Daily (QD) | Emraclidine 30 mg, Once Daily (QD)
Started | 128 | 128 | 129
Completed | 85 | 89 | 92
Not Completed | 43 | 39 | 37
Not completed — Adverse Event | 5 | 6 | 10
Not completed — Lack of Efficacy | 2 | 4 | 1
Not completed — Physician Decision | 6 | 0 | 4
Not completed — Withdrawal of consent | 28 | 27 | 21
Not completed — Other, not specified | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: all randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Emraclidine 10 mg, Once Daily (QD) | Emraclidine 30 mg, Once Daily (QD) | Total
Number analyzed (Participants) | 128 | 128 | 129 | 385
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (11.46) | 40.6 (11.28) | 42.5 (12.23) | 42.0 (11.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 31 | 27 | 89
  Male | 97 | 97 | 102 | 296
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 20 | 9 | 50
  Not Hispanic or Latino | 107 | 105 | 118 | 330
  Unknown or Not Reported | 0 | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 3 | 3
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 89 | 88 | 87 | 264
  White | 37 | 39 | 33 | 109
  More than one race | 2 | 1 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Week 6 in the Positive and Negative Syndrome Scale (PANSS) Total Score
Description: The PANSS measures symptom severity of participants with schizophrenia and contains 7 positive symptom scales, 7 negative system scales, and 16 general psychopathology symptom scales. Participants are rated from 1 to 7 on each symptom scale with a total minimum score of 30 and a maximum score of 210. A decrease in PANSS total score correlates with an improvement in schizophrenia symptoms.
Time Frame: Baseline through Week 6
Population: Modified Intent-to-Treat population (mITT): All randomized participants who received at least 1 dose of investigational medicinal product (IMP) and have both a Baseline and at least 1 post-Baseline PANSS assessment; participants with available data
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Emraclidine 10 mg, Once Daily (QD) | Emraclidine 30 mg, Once Daily (QD)
Number analyzed (Participants) | 87 | 90 | 93
units on a scale | -13.5 [-17.0 to -10.0] | -14.7 [-18.1 to -11.2] | -16.5 [-20.0 to -13.1]
Statistical Analysis 1: Comparison: Placebo vs Emraclidine 30 mg, Once Daily (QD); Emraclidine 30 mg versus Placebo; Test type: Superiority — Least-squares mean difference from Placebo and CIs were estimated using a mixed effects repeated measures model with fixed effects for treatment group, geographic region, visit, and treatment-by-visit interaction and Baseline value as a covariate. Participant was included as a random effect. An unstructured covariance structure was used; p = 0.1765, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -3.0, 95% CI 2-sided [-7.5 to 1.4], Standard Error of Mean 2.24 — Emraclidine 30 mg - Placebo
Statistical Analysis 2: Comparison: Placebo vs Emraclidine 10 mg, Once Daily (QD); Emraclidine 10 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.6007, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -1.2, 95% CI 2-sided [-5.6 to 3.3], Standard Error of Mean 2.26 — Emraclidine 10 mg - Placebo

2. Secondary Outcome: Change From Baseline at Week 6 in the Clinical Global Impression - Severity (CGI-S Score)
Description: The CGI-S captures clinician's response to: "Considering your total clinical experience, how mentally ill is the participant at this time?" The clinician's answer was based on the following scale: 0 = not assessed; 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; 7 = among the most extremely ill participants. Negative changes from Baseline indicate less mental illness.
Time Frame: Baseline through Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Emraclidine 10 mg, Once Daily (QD) | Emraclidine 30 mg, Once Daily (QD)
Number analyzed (Participants) | 87 | 90 | 93
units on a scale | -0.70 [-0.89 to -0.51] | -0.75 [-0.94 to -0.56] | -0.84 [-1.03 to -0.65]
Statistical Analysis 1: Comparison: Placebo vs Emraclidine 30 mg, Once Daily (QD); Emraclidine 30 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.2534, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.14, 95% CI 2-sided [-0.39 to 0.10], Standard Error of Mean 0.124 — Emraclidine 30 mg - Placebo
Statistical Analysis 2: Comparison: Placebo vs Emraclidine 10 mg, Once Daily (QD); Emraclidine 10 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.6774, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.05, 95% CI 2-sided [-0.30 to 0.19], Standard Error of Mean 0.125 — Emraclidine 10 mg - Placebo

3. Secondary Outcome: Change From Baseline at All Time Points in Positive and Negative Syndrome Scale (PANSS) Total Score
Description: as for outcome 1
Time Frame: Baseline; Weeks 1, 2, 3, 4, 5, and 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Emraclidine 10 mg, Once Daily (QD) | Emraclidine 30 mg, Once Daily (QD)
Number analyzed (Participants) | 127 | 124 | 127
units on a scale
  Week 1 | -5.2 [-7.3 to -3.0] | -5.7 [-7.8 to -3.6] | -6.2 [-8.3 to -4.1]
  Week 2: number analyzed (Participants) | 113 | 114 | 118
  Week 2 | -8.7 [-11.3 to -6.1] | -8.8 [-11.4 to -6.3] | -9.0 [-11.6 to -6.5]
  Week 3: number analyzed (Participants) | 108 | 106 | 110
  Week 3 | -10.3 [-13.1 to -7.5] | -10.0 [-12.8 to -7.2] | -11.3 [-14.1 to -8.6]
  Week 4: number analyzed (Participants) | 99 | 102 | 104
  Week 4 | -12.1 [-15.3 to -9.0] | -12.8 [-15.9 to -9.6] | -13.3 [-16.4 to -10.2]
  Week 5: number analyzed (Participants) | 93 | 96 | 97
  Week 5 | -13.2 [-16.5 to -9.9] | -14.0 [-17.3 to -10.7] | -14.7 [-18.0 to -11.4]
  Week 6: number analyzed (Participants) | 87 | 90 | 93
  Week 6 | -13.5 [-17.0 to -10.0] | -14.7 [-18.1 to -11.2] | -16.5 [-20.0 to -13.1]
Statistical Analysis 1: Comparison: Placebo vs Emraclidine 30 mg, Once Daily (QD); Week 1-- Emraclidine 30 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.3596, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -1.0, 95% CI 2-sided [-3.2 to 1.2], Standard Error of Mean 1.10 — Emraclidine 30 mg - Placebo
Statistical Analysis 2: Comparison: Placebo vs Emraclidine 10 mg, Once Daily (QD); Week 1-- Emraclidine 10 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.6053, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.6, 95% CI 2-sided [-2.7 to 1.6], Standard Error of Mean 1.10 — Emraclidine 10 mg - Placebo
Statistical Analysis 3: Comparison: Placebo vs Emraclidine 30 mg, Once Daily (QD); Week 2-- Emraclidine 30 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.8149, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.4, 95% CI 2-sided [-3.4 to 2.7], Standard Error of Mean 1.54 — Emraclidine 30 mg - Placebo
Statistical Analysis 4: Comparison: Placebo vs Emraclidine 10 mg, Once Daily (QD); Week 2-- Emraclidine 10 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.9058, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.2, 95% CI 2-sided [-3.2 to 2.9], Standard Error of Mean 1.55 — Emraclidine 10 mg - Placebo
Statistical Analysis 5: Comparison: Placebo vs Emraclidine 30 mg, Once Daily (QD); Week 3-- Emraclidine 30 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.5419, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -1.0, 95% CI 2-sided [-4.4 to 2.3], Standard Error of Mean 1.71 — Emraclidine 30 mg - Placebo
Statistical Analysis 6: Comparison: Placebo vs Emraclidine 10 mg, Once Daily (QD); Week 3-- Emraclidine 10 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.8585, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = 0.3, 95% CI 2-sided [-3.1 to 3.7], Standard Error of Mean 1.72 — Emraclidine 10 mg - Placebo
Statistical Analysis 7: Comparison: Placebo vs Emraclidine 30 mg, Once Daily (QD); Week 4-- Emraclidine 30 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.5521, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -1.2, 95% CI 2-sided [-5.1 to 2.7], Standard Error of Mean 1.99 — Emraclidine 30 mg - Placebo
Statistical Analysis 8: Comparison: Placebo vs Emraclidine 10 mg, Once Daily (QD); Week 4-- Emraclidine 10 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.7540, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.6, 95% CI 2-sided [-4.6 to 3.3], Standard Error of Mean 2.00 — Emraclidine 10 mg - Placebo
Statistical Analysis 9: Comparison: Placebo vs Emraclidine 30 mg, Once Daily (QD); Week 5-- Emraclidine 30 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.4842, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -1.5, 95% CI 2-sided [-5.7 to 2.7], Standard Error of Mean 2.12 — Emraclidine 30 mg - Placebo
Statistical Analysis 10: Comparison: Placebo vs Emraclidine 10 mg, Once Daily (QD); Week 5-- Emraclidine 10 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.6999, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.8, 95% CI 2-sided [-5.0 to 3.4], Standard Error of Mean 2.13 — Emraclidine 10 mg - Placebo
Statistical Analysis 11: Comparison: Placebo vs Emraclidine 30 mg, Once Daily (QD); Week 6-- Emraclidine 30 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.1765, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -3.0, 95% CI 2-sided [-7.5 to 1.4], Standard Error of Mean 2.24 — Emraclidine 30 mg - Placebo
Statistical Analysis 12: Comparison: Placebo vs Emraclidine 10 mg, Once Daily (QD); Week 6-- Emraclidine 10 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.6007, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -1.2, 95% CI 2-sided [-5.6 to 3.3], Standard Error of Mean 2.26 — Emraclidine 10 mg - Placebo

4. Secondary Outcome: Change From Baseline at All Time Points in the Clinical Global Impression - Severity (CGI-S) Score
Description: as for outcome 2
Time Frame: Baseline; Weeks 1, 2, 3, 4, 5, and 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Emraclidine 10 mg, Once Daily (QD) | Emraclidine 30 mg, Once Daily (QD)
Number analyzed (Participants) | 127 | 124 | 127
units on a scale
  Week 1 | -0.18 [-0.29 to -0.06] | -0.17 [-0.29 to -0.05] | -0.21 [-0.32 to -0.09]
  Week 2: number analyzed (Participants) | 114 | 114 | 118
  Week 2 | -0.36 [-0.50 to -0.21] | -0.39 [-0.54 to -0.25] | -0.35 [-0.50 to -0.21]
  Week 3: number analyzed (Participants) | 108 | 107 | 110
  Week 3 | -0.48 [-0.64 to -0.32] | -0.42 [-0.58 to -0.26] | -0.52 [-0.67 to -0.36]
  Week 4: number analyzed (Participants) | 99 | 102 | 104
  Week 4 | -0.54 [-0.71 to -0.36] | -0.53 [-0.70 to -0.36] | -0.70 [-0.87 to -0.53]
  Week 5: number analyzed (Participants) | 92 | 96 | 97
  Week 5 | -0.67 [-0.85 to -0.49] | -0.64 [-0.82 to -0.46] | -0.74 [-0.92 to -0.56]
  Week 6: number analyzed (Participants) | 87 | 90 | 93
  Week 6 | -0.70 [-0.89 to -0.51] | -0.75 [-0.94 to -0.56] | -0.84 [-1.03 to -0.65]
Statistical Analysis 1: Comparison: Placebo vs Emraclidine 30 mg, Once Daily (QD); Week 1-- Emraclidine 30 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.5822, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.03, 95% CI 2-sided [-0.15 to 0.09], Standard Error of Mean 0.061 — Emraclidine 30 mg - Placebo
Statistical Analysis 2: Comparison: Placebo vs Emraclidine 10 mg, Once Daily (QD); Week 1-- Emraclidine 10 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.9244, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = 0.01, 95% CI 2-sided [-0.11 to 0.13], Standard Error of Mean 0.061 — Emraclidine 10 mg - Placebo
Statistical Analysis 3: Comparison: Placebo vs Emraclidine 30 mg, Once Daily (QD); Week 2-- Emraclidine 30 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.9348, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = 0.01, 95% CI 2-sided [-0.17 to 0.18], Standard Error of Mean 0.088 — Emraclidine 30 mg - Placebo
Statistical Analysis 4: Comparison: Placebo vs Emraclidine 10 mg, Once Daily (QD); Week 2-- Emraclidine 10 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.7160, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.03, 95% CI 2-sided [-0.21 to 0.14], Standard Error of Mean 0.089 — Emraclidine 10 mg - Placebo
Statistical Analysis 5: Comparison: Placebo vs Emraclidine 30 mg, Once Daily (QD); Week 3-- Emraclidine 30 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.6883, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.04, 95% CI 2-sided [-0.24 to 0.16], Standard Error of Mean 0.100 — Emraclidine 30 mg - Placebo
Statistical Analysis 6: Comparison: Placebo vs Emraclidine 10 mg, Once Daily (QD); Week 3-- Emraclidine 10 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.5973, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = 0.05, 95% CI 2-sided [-0.14 to 0.25], Standard Error of Mean 0.100 — Emraclidine 10 mg - Placebo
Statistical Analysis 7: Comparison: Placebo vs Emraclidine 30 mg, Once Daily (QD); Week 4-- Emraclidine 30 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.1392, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.16, 95% CI 2-sided [-0.38 to 0.05], Standard Error of Mean 0.110 — Emraclidine 30 mg - Placebo
Statistical Analysis 8: Comparison: Placebo vs Emraclidine 10 mg, Once Daily (QD); Week 4-- Emraclidine 10 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.9421, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = 0.01, 95% CI 2-sided [-0.21 to 0.23], Standard Error of Mean 0.111 — Emraclidine 10 mg - Placebo
Statistical Analysis 9: Comparison: Placebo vs Emraclidine 30 mg, Once Daily (QD); Week 5-- Emraclidine 30 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.5431, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.07, 95% CI 2-sided [-0.30 to 0.16], Standard Error of Mean 0.116 — Emraclidine 30 mg - Placebo
Statistical Analysis 10: Comparison: Placebo vs Emraclidine 10 mg, Once Daily (QD); Week 5-- Emraclidine 10 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.8160, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = 0.03, 95% CI 2-sided [-0.20 to 0.26], Standard Error of Mean 0.117 — Emraclidine 10 mg - Placebo
Statistical Analysis 11: Comparison: Placebo vs Emraclidine 30 mg, Once Daily (QD); Week 6-- Emraclidine 30 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.2534, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.14, 95% CI 2-sided [-0.39 to 0.10], Standard Error of Mean 0.124 — Emraclidine 30 mg - Placebo
Statistical Analysis 12: Comparison: Placebo vs Emraclidine 10 mg, Once Daily (QD); Week 6-- Emraclidine 10 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.6774, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.05, 95% CI 2-sided [-0.30 to 0.19], Standard Error of Mean 0.125 — Emraclidine 10 mg - Placebo

5. Secondary Outcome: Percentage of Responders at Week 6 (Responders Defined as ≥30% Reduction From Baseline in Positive and Negative Syndrome Scale [PANSS] Total Score)
Description: The PANSS measures symptom severity of participants with schizophrenia and contains 7 positive symptom scales, 7 negative system scales, and 16 general psychopathology symptom scales. Participants are rated from 1 to 7 on each symptom scale with a total minimum score of 30 and a maximum score of 210. A decrease in PANSS total score correlates with an improvement in schizophrenia symptoms. A PANSS responder is defined as a participant with at least a 30% decrease in PANSS total score compared to Baseline at Week 6 visit or the early termination visit. If a participant discontinued and did not have an early termination visit, the participant's last assessment was considered.
Time Frame: Baseline through Week 6
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Emraclidine 10 mg, Once Daily (QD) | Emraclidine 30 mg, Once Daily (QD)
Number analyzed (Participants) | 127 | 125 | 127
percentage of participants | 10.2 | 17.6 | 17.3
Statistical Analysis 1: Comparison: Placebo vs Emraclidine 30 mg, Once Daily (QD); Emraclidine 30 mg versus Placebo; Test type: Superiority — Odds ratio, 95% confidence interval, and p-value were from a logistic regression with treatment group, geographic region and Baseline value as a covariate; p = 0.0904, Regression, Logistic; Odds Ratio = 1.90, 95% CI 2-sided [0.90 to 3.99]
Statistical Analysis 2: Comparison: Placebo vs Emraclidine 10 mg, Once Daily (QD); Emraclidine 10 mg versus Placebo; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.0756, Regression, Logistic; Odds Ratio = 1.96, 95% CI 2-sided [0.93 to 4.13]

6. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Event (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study drug. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent adverse events/treatment-emergent serious adverse events (TEAEs/TESAEs) are defined as any event that began or worsened in severity on or after the first dose of study drug.
Time Frame: From first dose of study drug until 28 days following last dose of study drug (up to Week 10)
Population: Full analysis set: All randomized participants who received at least 1 dose of investigational medicinal product (IMP)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Emraclidine 10 mg, Once Daily (QD) | Emraclidine 30 mg, Once Daily (QD)
Number analyzed (Participants) | 128 | 128 | 129
Participants
  Any TEAE | 73 | 78 | 82
  TESAE | 2 | 4 | 1

7. Secondary Outcome: Number of Participants With Clinically Significant Changes in Electrocardiogram (ECGs)
Description: 12-lead electrocardiogram (ECG) recordings were obtained after the participant had been supine and at rest for at least 3 minutes.
Time Frame: Baseline; from first dose of study drug up to Week 6
Population: Full analysis set: All randomized participants who received at least 1 dose of investigational medicinal product (IMP)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Emraclidine 10 mg, Once Daily (QD) | Emraclidine 30 mg, Once Daily (QD)
Number analyzed (Participants) | 128 | 128 | 129
Participants
  QTcF value > 450 - 480 msec | 5 | 3 | 1
  QTcF value > 480 - 500 msec | 0 | 0 | 0
  QTcF value > 500 msec | 0 | 0 | 0
  QTcF increase from Baseline > 30 - 60 msec | 13 | 8 | 8
  QTcF increase from Baseline > 60 msec | 1 | 1 | 0

8. Secondary Outcome: Number of Participants With Clinically Significant Changes in Clinical Laboratory Assessments
Description: Clinical laboratory tests were performed at scheduled study visits, and the investigator recorded any clinically significant changes.
Time Frame: Baseline; from first dose of study drug up to Week 6
Population: Full analysis set: All randomized participants who received at least 1 dose of investigational medicinal product (IMP)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Emraclidine 10 mg, Once Daily (QD) | Emraclidine 30 mg, Once Daily (QD)
Number analyzed (Participants) | 128 | 128 | 129
Participants | 3 | 4 | 4

9. Secondary Outcome: Number of Participants With Clinically Significant Changes in Vital Sign Measurements
Description: Vital signs were obtained after the participant had been supine and at rest for 3 minutes and included temperature, systolic and diastolic blood pressure, respiratory rate, and heart rate. Participants' body weights were also measured and recorded.
Time Frame: Baseline; from first dose of study drug up to Week 6
Population: Full analysis set: All randomized participants who received at least 1 dose of investigational medicinal product (IMP)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Emraclidine 10 mg, Once Daily (QD) | Emraclidine 30 mg, Once Daily (QD)
Number analyzed (Participants) | 128 | 128 | 129
Participants
  Supine Systolic Blood Pressure < 90 mmHg | 0 | 0 | 0
  Supine Systolic Blood Pressure > 140 mmHg and ≤ 160 mmHg | 15 | 9 | 11
  Supine Systolic Blood Pressure > 160 mmHg and ≤ 200 mmHg | 0 | 0 | 1
  Supine Systolic Blood Pressure > 200 mmHg | 0 | 0 | 0
  Orthostatic Change in Systolic Blood Pressure ≥ 20 mmHg decrease | 4 | 2 | 5
  Supine Diastolic Blood Pressure < 50 mmHg | 0 | 0 | 0
  Supine Diastolic Blood Pressure > 90 mmHg and ≤ 100 mmHg | 10 | 9 | 19
  Supine Diastolic Blood Pressure > 100 mmHg and ≤ 120 mmHg | 0 | 0 | 3
  Supine Diastolic Blood Pressure > 120 mmHg | 0 | 0 | 0
  Orthostatic Change in Diastolic Blood Pressure ≥ 10 mmHg decrease | 9 | 7 | 14
  Supine Heart Rate < 50 bpm | 1 | 0 | 0
  Supine Heart Rate ≥ 50 bpm and < 60 bpm | 17 | 6 | 6
  Supine Heart Rate > 100 bpm and ≤ 120 bpm | 8 | 18 | 24
  Supine Heart Rate > 120 bpm | 0 | 0 | 3
  Temperature < 36 °C | 1 | 3 | 5
  Temperature > 38 °C | 1 | 0 | 0
  Respiratory Rate < 12 breaths/min | 0 | 0 | 0
  Respiratory Rate > 20 breaths/min | 3 | 5 | 6
  Body Weight ≥ 7% decrease | 1 | 1 | 1
  Body Weight ≥ 7% increase | 16 | 24 | 14

10. Secondary Outcome: Number of Participants With Clinically Significant Changes in Physical and Neurological Examination Results
Description: The number of participants with clinically significant changes in physical and neurological examination results was documented.
Time Frame: Baseline; from first dose of study drug up to Week 6
Population: Full analysis set: All randomized participants who received at least 1 dose of investigational medicinal product (IMP)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Emraclidine 10 mg, Once Daily (QD) | Emraclidine 30 mg, Once Daily (QD)
Number analyzed (Participants) | 128 | 128 | 129
Participants
  Clinically Significant Changes in Physical Examination | 1 | 1 | 3
  Clinically Significant Changes in Neurological Examination | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Suicide-Related Treatment-Emergent Events Assessed Using the Columbia Suicide-Severity Rating Scale (C-SSRS)
Description: The C-SSRS rates an individual's degree of suicidal ideation (SI) on a scale, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent." The scale identifies SI severity and intensity, which may be indicative of an individual's intent to commit suicide. C-SSRS SI severity subscale ranges from 0 (no SI) to 5 (active SI with plan and intent).
Time Frame: Baseline; from first dose of study drug up to Week 6
Population: Full analysis set: All randomized participants who received at least 1 dose of investigational medicinal product (IMP)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Emraclidine 10 mg, Once Daily (QD) | Emraclidine 30 mg, Once Daily (QD)
Number analyzed (Participants) | 128 | 128 | 129
Participants
  Treatment-Emergent Suicidal Ideation Compared to Recent History | 1 | 2 | 7
  Treatment-Emergent Serious Suicidal Ideation Compared to Recent History | 0 | 0 | 0
  Emergence of Serious Suicidal Ideation Compared to Recent History | 0 | 0 | 0
  Emergence of Suicidal Behavior Compared to all Prior History | 0 | 0 | 0

12. Secondary Outcome: Change From Baseline in Simpson Angus Scale (SAS) Total Score
Description: The SAS consists of a list of 10 symptoms of Parkinsonism. Each item is rated on a 5-point scale, with a score of 0 representing absence of symptoms and a score of 4 representing a severe condition. The SAS total score is the sum of the scores for all 10 items. Negative changes from Baseline indicate an improvement in symptoms.
Time Frame: Baseline; Weeks 3 and 6
Population: Full analysis set: All randomized participants who received at least 1 dose of investigational medicinal product (IMP); participants with available data
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Emraclidine 10 mg, Once Daily (QD) | Emraclidine 30 mg, Once Daily (QD)
Number analyzed (Participants) | 119 | 119 | 125
units on a scale
  Week 3 | 0.0 [-0.1 to 0.1] | 0.0 [0.0 to 0.1] | 0.1 [0.0 to 0.2]
  Week 6: number analyzed (Participants) | 89 | 90 | 95
  Week 6 | 0.0 [-0.1 to 0.1] | 0.0 [-0.1 to 0.1] | 0.0 [-0.1 to 0.1]
Statistical Analysis 1: Comparison: Placebo vs Emraclidine 30 mg, Once Daily (QD); Week 3-- Emraclidine 30 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.2418, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = 0.1, 95% CI 2-sided [0.0 to 0.2], Standard Error of Mean 0.05 — Emraclidine 30 mg - Placebo
Statistical Analysis 2: Comparison: Placebo vs Emraclidine 10 mg, Once Daily (QD); Week 3-- Emraclidine 10 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.5720, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = 0.0, 95% CI 2-sided [-0.1 to 0.1], Standard Error of Mean 0.05 — Emraclidine 10 mg - Placebo
Statistical Analysis 3: Comparison: Placebo vs Emraclidine 30 mg, Once Daily (QD); Week 6-- Emraclidine 30 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.7459, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = 0.0, 95% CI 2-sided [-0.1 to 0.1], Standard Error of Mean 0.06 — Emraclidine 30 mg - Placebo
Statistical Analysis 4: Comparison: Placebo vs Emraclidine 10 mg, Once Daily (QD); Week 6-- Emraclidine 10 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.6729, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = 0.0, 95% CI 2-sided [-0.1 to 0.1], Standard Error of Mean 0.06 — Emraclidine 10 mg - Placebo

13. Secondary Outcome: Change From Baseline in Abnormal Involuntary Movement Scale (AIMS) Movement Rating Score
Description: The Abnormal Involuntary Movement Scale assessment consists of 10 items describing symptoms of dyskinesia. Facial and oral movements (items 1-4), extremity movements (items 5 and 6), and trunk movements (item 7) are observed unobtrusively while the participant is at rest, and the investigator also makes global judgments on the participant's dyskinesias (items 8-10). Each item is rated on a 5-point scale, with a score of 0 representing absence of symptoms (for item 10, no awareness), and a score of 4 indicating a severe condition (for item 10, awareness, severe distress). In addition, the AIMS includes 2 yes/no questions that address the participant's dental status.
  The AIMS Movement Rating Score is defined as the sum of individual scores from items 1-7, ranging from 0 to 28. A lower score indicates less severe or absent abnormal movements. A negative change in the mean from Baseline indicates improvement in the severity of abnormal involuntary movements.
Time Frame: Baseline; Weeks 3 and 6
Population: as for outcome 12
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Emraclidine 10 mg, Once Daily (QD) | Emraclidine 30 mg, Once Daily (QD)
Number analyzed (Participants) | 119 | 119 | 125
units on a scale
  Week 3 | 0.0 [-0.1 to 0.1] | -0.1 [-0.2 to 0.0] | 0.1 [0.0 to 0.2]
  Week 6: number analyzed (Participants) | 89 | 90 | 95
  Week 6 | 0.0 [-0.1 to 0.1] | 0.0 [-0.1 to 0.1] | 0.0 [-0.1 to 0.1]
Statistical Analysis 1: Comparison: Placebo vs Emraclidine 30 mg, Once Daily (QD); Week 3-- Emraclidine 30 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.3783, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = 0.1, 95% CI 2-sided [-0.1 to 0.2], Standard Error of Mean 0.06 — Emraclidine 30 mg - Placebo
Statistical Analysis 2: Comparison: Placebo vs Emraclidine 10 mg, Once Daily (QD); Week 3-- Emraclidine 10 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.2242, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.1, 95% CI 2-sided [-0.2 to 0.0], Standard Error of Mean 0.06 — Emraclidine 10 mg - Placebo
Statistical Analysis 3: Comparison: Placebo vs Emraclidine 30 mg, Once Daily (QD); Week 6-- Emraclidine 30 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.8626, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = 0.0, 95% CI 2-sided [-0.1 to 0.1], Standard Error of Mean 0.05 — Emraclidine 30 mg - Placebo
Statistical Analysis 4: Comparison: Placebo vs Emraclidine 10 mg, Once Daily (QD); Week 6-- Emraclidine 10 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.6106, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = 0.0, 95% CI 2-sided [-0.1 to 0.1], Standard Error of Mean 0.05 — Emraclidine 10 mg - Placebo

14. Secondary Outcome: Change From Baseline in Barnes Akathisia Rating Scale (BARS) Global Clinical Evaluation Score
Description: The BARS consists of 4 items related to akathisia: The first 3 items are rated on a 4-point scale, with a score of 0 representing absence of symptoms and a score of 3 representing a severe condition. The global clinical evaluation is made on a 6-point scale, with a score of 0 representing absence of symptom and a score of 5 representing severe akathisia. Negative changes from Baseline indicate an improvement in symptoms.
Time Frame: Baseline; Weeks 3 and 6
Population: as for outcome 12
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Emraclidine 10 mg, Once Daily (QD) | Emraclidine 30 mg, Once Daily (QD)
Number analyzed (Participants) | 119 | 119 | 125
units on a scale
  Week 3 | 0.0 [-0.1 to 0.0] | 0.0 [0.0 to 0.1] | 0.0 [0.0 to 0.1]
  Week 6: number analyzed (Participants) | 89 | 90 | 95
  Week 6 | 0.0 [0.0 to 0.0] | 0.0 [-0.1 to 0.0] | 0.0 [0.0 to 0.0]
Statistical Analysis 1: Comparison: Placebo vs Emraclidine 30 mg, Once Daily (QD); Week 3-- Emraclidine 30 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.4219, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = 0.0, 95% CI 2-sided [0.0 to 0.1], Standard Error of Mean 0.03 — Emraclidine 30 mg - Placebo
Statistical Analysis 2: Comparison: Placebo vs Emraclidine 10 mg, Once Daily (QD); Week 3-- Emraclidine 10 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.3933, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = 0.0, 95% CI 2-sided [0.0 to 0.1], Standard Error of Mean 0.03 — Emraclidine 10 mg - Placebo
Statistical Analysis 3: Comparison: Placebo vs Emraclidine 30 mg, Once Daily (QD); Week 6-- Emraclidine 30 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.7366, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = 0.0, 95% CI 2-sided [0.0 to 0.0], Standard Error of Mean 0.02 — Emraclidine 30 mg - Placebo
Statistical Analysis 4: Comparison: Placebo vs Emraclidine 10 mg, Once Daily (QD); Week 6-- Emraclidine 10 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.4639, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = 0.0, 95% CI 2-sided [-0.1 to 0.0], Standard Error of Mean 0.02 — Emraclidine 10 mg - Placebo

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from the time informed consent was signed to the end of the study. The median time on follow-up was 81.5 days for the Placebo group, 77 days for the Emraclidine 10 mg group, and 80 days for the Emraclidine 30 mg group.
Arm/Group | Placebo | Emraclidine 10 mg, Once Daily (QD) | Emraclidine 30 mg, Once Daily (QD)
All-Cause Mortality (participants affected / at risk) | 0/128 | 0/128 | 0/129
Serious Adverse Events (participants affected / at risk) | 2/128 | 4/128 | 1/129
Other Adverse Events (participants affected / at risk) | 56/128 | 66/128 | 74/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=128) | Emraclidine 10 mg, Once Daily (QD) (N=128) | Emraclidine 30 mg, Once Daily (QD) (N=129)
DYSTONIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
AGGRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
AGITATION (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
SCHIZOPHRENIA (Psychiatric disorders) | 2 (3) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=128) | Emraclidine 10 mg, Once Daily (QD) (N=128) | Emraclidine 30 mg, Once Daily (QD) (N=129)
SINUS TACHYCARDIA (Cardiac disorders) | 1 (1) | 2 (2) | 6 (8)
ABDOMINAL PAIN (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 4 (4) | 3 (3) | 3 (3)
DRY MOUTH (Gastrointestinal disorders) | 3 (3) | 5 (5) | 12 (12)
DYSPEPSIA (Gastrointestinal disorders) | 4 (5) | 5 (5) | 10 (10)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 (2) | 3 (3) | 4 (5)
NAUSEA (Gastrointestinal disorders) | 2 (2) | 3 (4) | 6 (7)
TOOTHACHE (Gastrointestinal disorders) | 3 (3) | 1 (1) | 3 (3)
FATIGUE (General disorders) | 1 (1) | 0 (0) | 5 (5)
TOOTH ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 3 (4)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 3 (3) | 4 (4) | 3 (3)
BLOOD PRESSURE INCREASED (Investigations) | 0 (0) | 0 (0) | 4 (4)
WEIGHT INCREASED (Investigations) | 11 (11) | 22 (22) | 8 (8)
INCREASED APPETITE (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 5 (6)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (2) | 8 (8)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (5) | 1 (1)
DIZZINESS (Nervous system disorders) | 4 (4) | 1 (1) | 3 (4)
HEADACHE (Nervous system disorders) | 12 (14) | 18 (20) | 17 (18)
SOMNOLENCE (Nervous system disorders) | 6 (6) | 9 (11) | 9 (9)
AGITATION (Psychiatric disorders) | 4 (4) | 1 (1) | 5 (8)
ANXIETY (Psychiatric disorders) | 3 (3) | 1 (1) | 3 (3)
INSOMNIA (Psychiatric disorders) | 5 (5) | 6 (7) | 3 (3)
PSYCHOTIC DISORDER (Psychiatric disorders) | 4 (4) | 3 (3) | 2 (2)
SCHIZOPHRENIA (Psychiatric disorders) | 2 (2) | 1 (1) | 4 (4)
SUICIDAL IDEATION (Psychiatric disorders) | 1 (1) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/90/NCT05227690/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/90/NCT05227690/SAP_001.pdf